CLINICAL TRIAL: NCT06446544
Title: Functional Residual Capacity and Alveolar Recruitment in Single-lung Ventilation: a Randomized Study
Acronym: OLVEELV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/0383/HP
Record Dates: First submitted 2024-02-26; First posted 2024-06-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Lung Injury
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm monitoring of the VPFE with intraoperative alveolar recruitment maneuvers (Experimental): arm monitoring of the VPFE with intraoperative alveolar recruitment maneuvers
  Interventions: Procedure: VPFE monitoring with intraoperative alveolar recruitment maneuvers.
- VPFE monitoring arm without intraoperative alveolar recruitment maneuvers. (Placebo Comparator): VPFE monitoring arm without intraoperative alveolar recruitment maneuvers.
  Interventions: Procedure: VPFE monitoring with intraoperative alveolar recruitment maneuvers.

INTERVENTIONS:
Procedure: VPFE monitoring with intraoperative alveolar recruitment maneuvers. — VPFE monitoring with intraoperative alveolar recruitment maneuvers.
  Arms: arm monitoring of the VPFE with intraoperative alveolar recruitment maneuvers
Procedure: VPFE monitoring with intraoperative alveolar recruitment maneuvers. — VPFE monitoring with intraoperative alveolar recruitment maneuvers.
  Arms: VPFE monitoring arm without intraoperative alveolar recruitment maneuvers.

SUMMARY:
In thoracic surgery, the incidence of postoperative pulmonary complications is higher than for other surgeries. Indeed, thoracic surgery has the specificity of being carried out with single-lung ventilation and is thus a source of intraoperative atelectasis which persists postoperatively and gives rise to pulmonary complications, particularly infectious ones. During one-lung ventilation, mediastinal and abdominal compression on the ventilated lung leads to a drop in functional residual capacity (FRC) which will in turn lead to collapse of the small airways leading to the formation of atelectasis.

Strategies exist to limit the appearance of atelectasis. One of the intraoperative strategies is alveolar recruitment. Alveolar recruitment is a dynamic process that can be defined by a transient increase in transpulmonary pressure beyond the critical opening pressure. Physiologically, alveolar recruitment corresponds to the re-aeration of poorly or non-aerated lung areas. In single-lung ventilation, intraoperative alveolar recruitment maneuvers are not performed systematically to prevent the formation of atelectasis.

The General Electric Carescape R860 ventilator allows intraoperative monitoring of end-expiratory closing lung volume (EFVP), which corresponds to the CRF associated with positive expiratory pressure (PEEP). This spirometry incorporated in the ventilator continuously monitors the intraoperative variation of VPFE, thus making it possible to detect any significant decrease which would favor the formation of intraoperative atelectasis. Early detection of VPFE can therefore allow the anesthetist-resuscitator to initiate intraoperative alveolar recruitment maneuvers adapted to the patient. Alveolar recruitment maneuvers are then personalized and based on precise monitoring of the evolution of the VPFE.

The effectiveness of recruitment maneuvers can be evaluated and quantified (with the Lung Ultrasound Score (LUS)) postoperatively using pleuropulmonary ultrasound. Thus, early ultrasound detection, from the post-interventional monitoring room (SSPI), would make it possible to undertake rapid therapeutic maneuvers to combat the atelectasis observed. A patient could benefit, for example, from prophylactic NIV from the recovery room, from a stricter postural program in a seated position, or from an earlier and/or more intensive respiratory rehabilitation program with the physiotherapy team.

DETAILED DESCRIPTION:
In thoracic surgery, the incidence of postoperative pulmonary complications is higher than for other surgeries. Indeed, thoracic surgery has the specificity of being carried out with single-lung ventilation and is thus a source of intraoperative atelectasis which persists postoperatively and gives rise to pulmonary complications, particularly infectious ones. During one-lung ventilation, mediastinal and abdominal compression on the ventilated lung leads to a drop in functional residual capacity (FRC) which will in turn lead to collapse of the small airways leading to the formation of atelectasis.

Strategies exist to limit the appearance of atelectasis. One of the intraoperative strategies is alveolar recruitment. Alveolar recruitment is a dynamic process that can be defined by a transient increase in transpulmonary pressure beyond the critical opening pressure. Physiologically, alveolar recruitment corresponds to the re-aeration of poorly or non-aerated lung areas. In single-lung ventilation, intraoperative alveolar recruitment maneuvers are not performed systematically to prevent the formation of atelectasis.

The General Electric Carescape R860 ventilator allows intraoperative monitoring of end-expiratory closing lung volume (EFVP), which corresponds to the CRF associated with positive expiratory pressure (PEEP). This spirometry incorporated in the ventilator continuously monitors the intraoperative variation of VPFE, thus making it possible to detect any significant decrease which would favor the formation of intraoperative atelectasis. Early detection of VPFE can therefore allow the anesthetist-resuscitator to initiate intraoperative alveolar recruitment maneuvers adapted to the patient. Alveolar recruitment maneuvers are then personalized and based on precise monitoring of the evolution of the VPFE.

The effectiveness of recruitment maneuvers can be evaluated and quantified (with the Lung Ultrasound Score (LUS)) postoperatively using pleuropulmonary ultrasound. Thus, early ultrasound detection, from the post-interventional monitoring room (SSPI), would make it possible to undertake rapid therapeutic maneuvers to combat the atelectasis observed. A patient could benefit, for example, from prophylactic NIV from the recovery room, from a stricter postural program in a seated position, or from an earlier and/or more intensive respiratory rehabilitation program with the physiotherapy team.

ELIGIBILITY:
* Adult patient aged 18 to 75 years inclusive
* Patient requiring lobectomy or segmentectomy by video or robot-thoracoscopy
* Patient having read and understood the information letter and signed the consent form
* Patient affiliated to a social security system
* Women :

  * Of childbearing age (defined by the CTFG as a fertile woman, after menarche and until menopause, except in cases of permanent sterility (including hysterectomy, bilateral salpingectomy or bilateral oophorectomy))

    * using effective contraception according to the WHO (combined hormonal contraception (containing estrogens and progestins), progestin-only contraception, intrauterine device (IUD), male or female condoms) for at least 4 weeks before inclusion and during the study And,
    * Presenting a negative urine pregnancy test at inclusion;
  * Menopause: menopause according to the CTFG is defined as the absence of periods for 12 months without any other medical cause. An elevated follicle-stimulating hormone (FSH) level in the postmenopausal interval can be used to confirm a postmenopausal state in women who are not using hormonal contraception or hormone replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

Exclusion Criteria:

* Patients aged 76 and over
* COPD patients (Gold stage 3 or 4 of the 2023 Gold classification)
* Patients with a history of ischemic coronary artery disease
* Patients with a history of pulmonary emphysema bubbles on the ventilated lung
* Tracheostomized patient
* Obese patients (>30 kg/m²)
* Patients with a history of pulmonary resection
* ASA patients ≥4
* Patient benefiting from a pre-operative rehabilitation protocol with physiotherapy
* Pregnant or parturient or breastfeeding woman or proven absence of contraception
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection/under guardianship or curatorship
* History of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participation in the protocol or preventing them from giving informed consent
* Patient refusing to give consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of VPFE monitoring with intraoperative alveolar recruitment maneuvers compared to VPFE monitoring without intraoperative alveolar recruitment maneuvers on pulmonary aeration of the ventilated lung | 30 min post-extubation
  The primary endpoint will be the value of the LUS (Lung Ultrasound Score) score on the ventilated lung at the time of lung ultrasound in SSPI, 30 minutes after extubation (presence of atelectasis with a LUS score > or = 10/18).

IPD SHARING:
Plan to Share IPD: No